CLINICAL TRIAL: NCT03953079
Title: A Phase 2b Multicenter Dose-Ranging Study Evaluating the Safety and Efficacy of Sunitinib Malate Depot Formulation (GB-102) Compared to Aflibercept in Subjects With Neovascular (Wet) Age-related Macular Degeneration (ALTISSIMO Study)
Brief Title: A Depot Formulation of Sunitinib Malate (GB-102) Compared to Aflibercept in Subjects With Wet AMD
Acronym: ALTISSIMO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Graybug Vision (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GBV-102-002
Record Dates: First submitted 2019-05-13; First posted 2019-05-16 (Actual); Results first posted 2022-01-11 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Neovascular Age-Related Macular Degeneration
Keywords: Age-related macular degeneration (AMD); Choroidal neovascularization
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Sunitinib; aflibercept

STUDY DESIGN:
Intervention Model Description: Parallel-arm design
Who Masked: Outcomes Assessor
Masking Description: Visual examiner-masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- GB-102 1 mg/1 mg (Experimental): Participants will receive intravitreal (IVT) GB-102 1 mg in the study eye at Baseline and Month 6 and sham at Months 2, 4, 8 and 10.
  Interventions: Drug: Drug: GB-102
- GB-102 2 mg/1 mg (Experimental): Participants will receive intravitreal (IVT) GB-102 2 mg in the study eye at Baseline, intravitreal (IVT) GB-102 1 mg at Month 6 and sham at Months 2, 4, 8 and 10.
  Interventions: Drug: Drug: GB-102
- Aflibercept 2 mg (Active Comparator): Participants will receive intravitreal (IVT) aflibercept 2 mg in the study eye at Baseline, Months 2, 4, 6, 8 and 10.
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Drug: GB-102 — Intravitreal injection of GB-102
  Other Names: Sunitinib malate
  Arms: GB-102 1 mg/1 mg; GB-102 2 mg/1 mg
Drug: Aflibercept — Intravitreal injection of aflibercept (2 mg dose)
  Other Names: Eylea
  Arms: Aflibercept 2 mg

SUMMARY:
Phase 2b, multicenter, visual examiner-masked, randomized active-controlled, parallel-arm design study to evaluate the safety and duration of repeated IVT injections of 3 dose levels of GB-102 compared with aflibercept.

DETAILED DESCRIPTION:
Phase 2b, multicenter, visual examiner-masked, randomized active-controlled, parallel-arm design study to evaluate the safety and duration of the effect of GB-102, as measured by time to first rescue treatment across multiple dose levels of GB-102 administered every 6 months as compared to intravitreal (IVT) aflibercept administered every 2 months in subjects with neovascular (wet) age-related macular degeneration who have received prior induction with anti-vascular endothelial growth factor (VEGF)

Extension Study:

To monitor the safety and duration of effect of IVT GB-102 administered every 6 months compared to IVT aflibercept administered every 2 months in subjects in ALTISSIMO (Core Study) who complete all study visits through Month 12 (Day 360) and who do not require/receive rescue treatment at the Month 12 (Day 360) final study visit

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥ 50 years of age
* Presence of a choroidal neovascularization (CNV) lesion secondary to AMD treated with at least 3 prior intravitreal (IVT) injections of an anti-vascular endothelial growth factor (VEGF) agent (aflibercept, bevacizumab, or ranibizumab).
* Demonstrated response to prior anti-VEGF treatment since diagnosis
* Best-corrected visual acuity (BCVA) of 35 letters or better

Exclusion Criteria:

* History, within 6 months prior to screening, of any of the following: myocardial infarction, any cardiac event requiring hospitalization, treatment for acute congestive heart failure, transient ischemic attack, or stroke
* Uncontrolled hypertension, diabetes mellitus or intraocular pressure (IOP)
* Chronic renal disease
* Abnormal liver function
* Women who are pregnant or lactating

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Graybug Vision, Inc.
Locations (33):
- United States (33):
  - Retinal Consultants AZ, Gilbert, Arizona
  - Retinal Research Institute, Phoenix, Arizona
  - California Retina Research Consultants, Bakersfield, California
  - Retinal Diagnostic Center of Northern California, Campbell, California
  - The Retina Partners, Encino, California
  - Retina Consultants of Orange County, Fullerton, California
  - Northern California Retina Vitreous Associates Medical Group, Inc., Mountain View, California
  - West Coast Retina Medical Group, Inc., San Francisco, California
  - California Retina Consultants - CRC, Santa Barbara, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Specialty Retina Center, Coral Springs, Florida
  - Florida Retina Institute, Orlando, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Eye Associates of Pinellas, Pinellas Park, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Retina Consultants of Hawaii, ‘Aiea, Hawaii
  - University Retina and Macula, Lemont, Illinois
  - Wolfe Eye Clinic - West Des Moines, Des Moines, Iowa
  - Eye Associates of Northeast Louisiana, West Monroe, Louisiana
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Mid Atlantic Retina Specialists, Hagerstown, Maryland
  - Sierra Eye Associates, Reno, Nevada
  - Ophthalmic Consultants of Long Island, Oceanside, New York
  - Sterling Research, Cincinnati, Ohio
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Retina Research Institute of Texas, Abilene, Texas
  - Austin Retina Associates, Austin, Texas
  - Retina Research Center, PLLC, Austin, Texas
  - Retina Specialists, Plano, Texas
  - Retina Consultants of Houston, The Woodlands, Texas
  - Strategic Clinical Research Group LLC, Willow Park, Texas
  - Piedmont Eye Center, Lynchburg, Virginia
  - Retina Center NW PLLC, Silverdale, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- GB-102 1 mg/1 mg: Participants receive intravitreal (IVT) GB-102 1 mg in the study eye at Baseline and Month 6 and sham at Months 2, 4, 8 and 10.
- GB-102 2 mg/1 mg: Participants receive intravitreal (IVT) GB-102 2 mg in the study eye at Baseline, intravitreal (IVT) GB-102 1 mg at Month 6 and sham at Months 2, 4, 8 and 10.
- Aflibercept 2 mg: Participants receive intravitreal (IVT) aflibercept 2 mg in the study eye at Baseline, Months 2, 4, 6, 8 and 10.
Period: Core Study
Arm/Group | GB-102 1 mg/1 mg | GB-102 2 mg/1 mg | Aflibercept 2 mg
Started | 21 | 22 | 13
Completed | 20 | 18 | 12
Not Completed | 1 | 4 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 1
Not completed — COVID-19 | 0 | 1 | 0
Not completed — Difficulties leaving the house | 0 | 1 | 0
Period: Extension Study
Arm/Group | GB-102 1 mg/1 mg | GB-102 2 mg/1 mg | Aflibercept 2 mg
Started | 12 | 10 | 6
Completed (Completed Month 18 without receiving a rescue treatment.) | 6 | 4 | 1
Not Completed | 6 | 6 | 5
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Received Rescue Treatment | 5 | 6 | 5

BASELINE CHARACTERISTICS:
Population: Safety Set includes all subjects all randomized subjects who receive at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | GB-102 1 mg/1 mg | GB-102 2 mg/1 mg | Aflibercept 2 mg | Total
Number analyzed (Participants) | 21 | 22 | 13 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1 | 2
  >=65 years | 21 | 21 | 12 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 80 (8.08) | 77.8 (8.58) | 77.5 (9.13) | 78.5 (8.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 8 | 36
  Male | 6 | 9 | 5 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 20 | 22 | 13 | 55
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 20 | 22 | 12 | 54
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 22 | 13 | 56
Best Corrected Visual Acuity (ETDRS Letters) [Mean (Standard Deviation); unit: ETDRS letters] — Best corrected visual acuity (BCVA) measured using the Early Treatment of Diabetic Retinopathy Study (ETDRS) letters.
  BCVA ETDRS letters range from 0 (worst) to 100 (best)
  ETDRS letters | 70.8 (11.50) | 70.7 (9.92) | 69.6 (14.67) | 70.5 (11.52)
Central Subfield Thickness [Mean (Standard Deviation); unit: microns] | 211.0 (47.14) | 232.5 (54.37) | 217.5 (31.66) | 221.0 (47.42)

OUTCOME MEASURES:

1. Primary Outcome: Time to First Rescue Treatment
Description: Kaplan-Meier estimate of the median time to first rescue treatment.
Time Frame: Baseline through 12 months
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | GB-102 1 mg/1 mg | GB-102 2 mg/1 mg | Aflibercept 2 mg
Number analyzed (Participants) | 21 | 22 | 13
months | 5 [3 to 8] | 4 [3 to 4] | NA [NA to NA] — NA = not applicable/ not estimable due to small sample size and insufficient number of participants who needed rescue treatment.

2. Secondary Outcome: Time to Fulfillment of at Least One Rescue Criterion
Description: Assessment of time to fulfillment of at least one rescue criterion starting at the Month 6 visit through to the Month 12 visit
Time Frame: 6 months through 12 months
Population: Full Analysis Set which include all randomized subjects who received at least one dose of study treatment and complete a baseline and at least one post-baseline visit.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | GB-102 1 mg/1 mg | GB-102 2 mg/1 mg | Aflibercept 2 mg
Number analyzed (Participants) | 16 | 14 | 12
months | 1.5 [1 to 2] | 2 [NA to NA] — NA = not applicable/ not estimable due to small sample size and insufficient number of participants who met rescue criteria. | NA [6 to NA] — NA = not applicable/ not estimable due to small sample size and insufficient number of participants who met rescue criteria.

3. Secondary Outcome: Number of Times That at Least One Rescue Criterion is Met
Description: Assessment of the number of monthly intervals that at least one rescue criterion is met
Time Frame: Baseline through 12 months
Population: The Full Analysis Set (FAS) will include all randomized subjects who receive at least one dose of study treatment, and complete a baseline and at least one post-baseline visit.
Measure: Mean (Standard Error); unit: total monthly interval
Arm/Group | GB-102 1 mg/1 mg | GB-102 2 mg/1 mg | Aflibercept 2 mg
Number analyzed (Participants) | 21 | 22 | 13
total monthly interval | 5.1 (3.38) | 6.1 (2.86) | 1.1 (1.26)

4. Secondary Outcome: Number of Treatments, Including Both Rescue and Scheduled Study Treatments, During the Study
Description: Assessment of the number of treatments, including both rescue and scheduled study treatments, that occurred during the study
Time Frame: Baseline through 12 months
Population: as for outcome 3
Measure: Median (Full Range); unit: Injections
Arm/Group | GB-102 1 mg/1 mg | GB-102 2 mg/1 mg | Aflibercept 2 mg
Number analyzed (Participants) | 21 | 22 | 13
Injections | 4 [1 to 8] | 4 [1 to 7] | 6 [3 to 7]

5. Secondary Outcome: Change From Baseline in Best-corrected Visual Acuity (BCVA) (ETDRS Letter Score) at All Visits
Description: BCVA = best corrected visual acuity; ETDRS = early treatment of diabetic retinopathy
  BCVA ETDRS range = 0 (worst) to 100 (best)
  Assessment of change in BCVA (ETDRS letter score) from baseline at all visits
Time Frame: Baseline through 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: letters
Groups:
- Dose: Participants receive intravitreal (IVT) aflibercept 2 mg in the study eye at Baseline, Months 2, 4, 6, 8 and 10.
Arm/Group | GB-102 1 mg/1 mg | GB-102 2 mg/1 mg | Dose
Number analyzed (Participants) | 20 | 18 | 12
letters | -7.4 (4.72) | -5.1 (4.37) | 1.8 (0.97)

6. Secondary Outcome: Categorical Change From Baseline in BCVA (ETDRS Letter Score) at All Visits
Description: BCVA = best corrected visual acuity; ETDRS = early treatment of diabetic retinopathy
  BCVA ETDRS range = 0 (worst) to 100 (best)
  Assessment of categorical change in BCVA (ETDRS letter score) from baseline at all visits
Time Frame: Baseline through 12 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GB-102 1 mg/1 mg | GB-102 2 mg/1 mg | Aflibercept 2 mg
Number analyzed (Participants) | 20 | 18 | 12
Participants
  <= -15 letters | 7 | 4 | 0
  >= -14 to <= -10 letters | 3 | 2 | 2
  >= -9 to <= -5 letters | 1 | 1 | 1
  >= -4 to <= 4 letters | 7 | 8 | 5
  >= 5 to <= 9 letters | 2 | 2 | 3
  >= 10 to <= 14 letters | 0 | 1 | 1
  >= 15 letters | 0 | 0 | 0

7. Secondary Outcome: Frequency of Subjects With BCVA Worse Than 20/200 (Snellen Equivalent) at All Visits
Description: Assessment of the frequency of subjects with BCVA worse than 20/200 (Snellen equivalent) at all visits
  A vision score of 20/20 is considered normal. A vision score of 20/200 is considered legally blind.
Time Frame: Baseline through 12 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GB-102 1 mg/1 mg | GB-102 2 mg/1 mg | Aflibercept 2 mg
Number analyzed (Participants) | 20 | 18 | 12
Participants | 3 | 1 | 0

8. Secondary Outcome: Change From Baseline in Central Subfield Thickness (CST) (μm) at All Visits
Description: CST = central subfield thickness
  Assessment of change in CST (μm) measurement from baseline at all visits
Time Frame: Baseline through 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | GB-102 1 mg/1 mg | GB-102 2 mg/1 mg | Aflibercept 2 mg
Number analyzed (Participants) | 20 | 18 | 12
microns | 41.7 (20.69) | 27.2 (11.07) | 7.8 (15.46)

9. Secondary Outcome: Frequency of Subjects With Absence of Exudation (Intra-/Sub-retinal Fluid/Cystoid Edema) at at All Visits
Description: Assessment of the frequency of subjects with absence of exudation (intra-/sub-retinal fluid/cystoid edema) at all visits
Time Frame: Baseline through 12 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GB-102 1 mg/1 mg | GB-102 2 mg/1 mg | Aflibercept 2 mg
Number analyzed (Participants) | 16 | 16 | 9
Participants | 2 | 3 | 1

ADVERSE EVENTS:
Time Frame: Baseline to Month 18
Arm/Group | GB-102 1 mg/1 mg | GB-102 2 mg/1 mg | Aflibercept 2 mg
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22 | 0/13
Serious Adverse Events (participants affected / at risk) | 2/21 | 4/22 | 1/13
Other Adverse Events (participants affected / at risk) | 20/21 | 22/22 | 8/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GB-102 1 mg/1 mg (N=21) | GB-102 2 mg/1 mg (N=22) | Aflibercept 2 mg (N=13)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acute myeloid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GB-102 1 mg/1 mg (N=21) | GB-102 2 mg/1 mg (N=22) | Aflibercept 2 mg (N=13)
Vitreous floaters (Eye disorders) | 6 (8) | 10 (13) | 2 (2)
Iritis (Eye disorders) | 5 (6) | 10 (11) | 0 (0)
Retinal haemorrhage (Eye disorders) | 4 (4) | 4 (4) | 1 (1)
Visual acuity reduced (Eye disorders) | 3 (4) | 4 (4) | 0 (0)
Subretinal fluid (Eye disorders) | 2 (2) | 2 (2) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 5 (6) | 1 (1)
Cataract (Eye disorders) | 2 (4) | 3 (3) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 2 (3) | 0 (0)
Posterior capsule opacification (Eye disorders) | 1 (1) | 1 (1) | 1 (2)
Vitritis (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Subretinal fibrosis (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal thickening (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Vitreous detachment (Eye disorders) | 1 (2) | 0 (0) | 1 (2)
Episcleritis (Eye disorders) | 0 (0) | 3 (3) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 2 (2) | 1 (2)
Anterior chamber inflammation (Eye disorders) | 0 (0) | 2 (3) | 0 (0)
Cataract subcapsular (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Corneal oedema (Eye disorders) | 0 (0) | 2 (3) | 0 (0)
Keratic precipitates (Eye disorders) | 0 (0) | 2 (4) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 2 (3) | 0 (0)
Choroidal neovascularisation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatochalasis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye allergy (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Iris adhesions (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Papilloedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Punctate keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Scleritis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vitreous degeneration (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Neovascular age-related macular degeneration (Eye disorders) | 0 (0) | 1 (1) | 2 (3)
Subretinal hyperreflective exudation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Product residue present (Investigations) | 4 (4) | 6 (7) | 0 (0)
Intraocular pressure increased (Investigations) | 1 (1) | 1 (4) | 0 (0)
Optical coherence tomography abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Asymptomatic COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gingival abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Loose tooth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal wall neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Lens discolouration (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dry age-related macular degeneration (Eye disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Small sample size hinders the ability to compare groups statistically.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any investigator wishing to publish or present any study finding must present a manuscript or abstract to Graybug Vision 120 days prior to submission for publication or presentation to provide Graybug Vision an opportunity for review and comment.

DOCUMENTS (2):
  • Study Protocol (2020-09-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT03953079/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT03953079/SAP_001.pdf